CLINICAL TRIAL: NCT03927053
Title: Consequences of Marijuana Use on Inflammatory Pathways in HIV-Infected Youth
Brief Title: Consequences of Marijuana Use in HIV-infected Youth
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00100780
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Youth With HIV
Keywords: substance use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma biomarker measurements, toxicology measurements, proteomics studies, transcriptome analyses, flow cytometric analysis and storage. Cryopreserved peripheral blood cells, serum and plasma .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HIV infected youth who use marijuana only
- HIV infected youth who use tobacco only
- HIV infected youth who use tobacco and marijuana
- HIV infected youth with no substance use

SUMMARY:
Proposed study focuses on Youth With HIV (YWH) recruited from the University of North Carolina using a cross sectional assessment of blood samples, clinical, demographic, behavioral, [including substance use and frequency], and neurocognitive data will be evaluated from YWH treated before CD4 T cell decline.

DETAILED DESCRIPTION:
The long-term goal for the proposed research is to apply a systems biology approach to discover evidence that provides the basis for understanding the complex and at times conflicting roles for marijuana in chronic inflammation in HIV-infected youth. To achieve the goal, a systems biology approach with two aims is designed:

Aim 1. To identify inflammatory immune pathways perturbed by recreational marijuana with or without concomitant use of tobacco products by applying a deep sequencing approach to define global transcriptome of peripheral blood cells from HIV-infected virally suppressed youth.

Aim 2. To develop biomarker profiles associated with pro- or anti-inflammatory pathways perturbed by marijuana and to discover biomarker profiles linked to neurocognitive impairment that are impacted by marijuana and tobacco use by YWH

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years 0 days - less than28 years 364 days
* Currently treated with stable ART and no ART changes for >6months.
* Willingness to participate in CASI questionnaire of self-reported substance use
* Documented behavioral transmission of HIV infection based on CLIA approved HIV antibody/antigen based testing method in medical record -HIV diagnosis greater than or equal to years. Viral load LESS THAN 50 COPIES/ML for the past 6 months. --

Patients may have had single blips in viral load to greater than 50 but less than 1000 copies/ml within the year prior to screening.

* Current Substance profile by chart review or phone screening:
* Marijuana use defined as marijuana use by any route at least 3 times per week in the absence of tobacco. N= 20.
* Tobacco use only based on report of regular (at least 3 times per week smoking). N=24
* Tobacco plus marijuana use defined as regular smoking and marijuana (at least 3 times per week) N =7
* No substance use of any type (alcohol, tobacco, marijuana or other recreational drugs in the past 90 days). N = 10
* Able to provide written informed consent in English and to adhere to protocol schedule

Exclusion Criteria:

* History of AIDS defining illness
* Pregnancy at any time during the study
* Use of substances that would interfere with the ability to complete the study
* History of significant cognitive or motor impairment or other chronic condition that would interfere with the ability to complete the study and impact neurocognitive testing
* Acute psychiatric symptoms (e.g. suicidality, mania, psychosis or severe depression)
* Other neurological disorder (e.g. multiple sclerosis, seizure disorder, etc.) requiring ongoing treatment or active outpatient evaluation
* Severe mental illness (requiring antipsychotic or mood stabilizing medications and/or inpatient hospitalization in past year)
* History of CNS infection (AIDS opportunistic (e.g. toxoplasmosis) or non-opportunistic (bacterial meningitis) with lasting or permanent neurological sequelae)
* Underlying and/or uncontrolled medical illnesses that may result in chronic inflammation , (e.g. SLE or autoimmune disease) as determined by the PI
* Nursing mothers
* Unable to read and write in English

Ages: 21 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Enrollment will consist of approximately 61 HIV-infected youth meeting the below entry criteria who are receiving antiretroviral therapy with undetectable viral levels at the time of entry (based on viral load assay within 1 year of enrollment) Recruitment will include Youth Age 21-28
  * Youth who use marijuana only [targeted number 20 participants]
  * Youth who use tobacco products only [targeted number 24 participants]
  * Youth who use marijuana and tobacco [targeted number 7 participants]
  * Youth who do not use substances [targeted number 10 participants]
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Number of bio-marker pathways that are abnormal. | 24 months
  This is measured by molecular mechanism of chronic macrophage activation.
Plasma levels of sCD163 | 24 months
  Chi-square test will be used to compare discrete variables
Neurocognitive function as measured by Trial Making Test (TMT) | 24 months
Neurocognitive function as measured by WAIS-III (5 subtest IQ estimate) | 24 months
Neurocognitive function as measured by Hopkins Verbal Learning Test-R | 24 months
Neurocognitive function as measured by the Brief Visuospatial Memory Test-R | 24 months
Neurocognitive function as measured by the WRAT-4 Word Reading subtest | 24 months
Neurocognitive function as measured by Activities of Daily Living Questionnaire | 24 months
Neurocognitive function as measured by Behavior Rating Inventory of Executive Functioning | 24 months
Neurocognitive function as measured by Grooved Pegboard test | 24 months
Neurocognitive function as measured by Timed Gait Test | 24 months
Neurocognitive function as measured by Verbal Fluency Test | 24 Months
Neurocognitive function as measured by Brief Symptom Inventory | 24 months
Neurocognitive function as measured by Beck Depression Inventory-II | 24 months
Neurocognitive function as measured by ASSIST (substance abuse) | 24 months
Neurocognitive function as measured by Base ATN Adherence Questions | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: John W sleasman, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke UMC, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No